CLINICAL TRIAL: NCT01587378
Title: A Prospective, Randomized, Double-blind, Multi-centre Study, Where the Possible Effect of Metformin to Prevent Late Miscarriage and Preterm Delivery is Studied in Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: Metformin to Prevent Late Miscarriage and Preterm Delivery in Women With Polycystic Ovary Syndrome
Acronym: PregMet2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Vestre Viken Hospital Trust (Other); Landspitali University Hospital (Other); Uppsala University Hospital (Other); Haukeland University Hospital (Other); Karolinska University Hospital (Other); St. Olavs Hospital (Other); Sykehuset Telemark (Other Government); Alesund Hospital (Other); The Hospital of Vestfold (Other); Nordlandssykehuset HF (Other); Norrlands universitetssjukhus Umeå (Unknown); Sykehuset Innlandet HF (Other); Vestre Viken Ringerike Sykehus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011/1434; 2011-002203-15 (EudraCT Number)
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy; Polycystic Ovary Syndrome
Keywords: miscarriage; preterm birth; prevention
MeSH Terms: conditions — Polycystic Ovary Syndrome; Abortion, Spontaneous; Premature Birth | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metformin (Experimental)
  Interventions: Drug: Metformin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Metformin — Metformin 500 mg tablets, 1 tablet x 2 daily the first week and then 2 tablets x 2 daily from the second week to delivery
  Arms: metformin
Drug: placebo — identical placebo tablets, 1 tablet x 2 daily the first week and then 2 tablets x 2 daily from the second week to delivery
  Arms: placebo

SUMMARY:
The overall aim of the PregMet 2 Study is to investigate whether metformin prevents late miscarriages and preterm deliveries in PCOS women treated with metformin from first trimester of pregnancy to delivery in a large, randomized, controlled, multi-centre trial setting.

The investigators hypothesis is that metformin compared to placebo treatment from the first trimester to term, reduces the prevalence of late miscarriage (gestational week 13-22) and preterm birth (gestational week < 37) in PCOS women diagnosed according to Rotterdam 2003 consensus criteria, with singleton pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 years
* PCOS diagnosed or reconfirmed according to Rotterdam 2003 criteria, not more than 5 years prior to inclusion
* Mode of conception: Any
* Single, viable fetus, diagnosed by vaginal ultrasound
* Gestational week at inclusion: week 6 + 0 to 12 + 0
* Wash out for metformin: at least 7 days
* Able to communicate fluently in the official language at the study cite or English

Exclusion Criteria:

* Any type of diabetes (except GDM in former pregnancy)
* Known liver disease or ALAT > 100 IU/L
* Known kidney disease or creatinine > 110 μmol/L
* Known alcohol or drug abuse
* Use of drugs interfering with metformin: erytromycin (or other macrolides), cimetidine, anticoagulation therapy
* Unsuitable for participation of other reasons

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 489 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
combined incidence of late miscarriages and preterm births | at delivery
  This includes spontaneous births, induced vaginal deliveries and operative deliveries on medical indications.

SECONDARY OUTCOMES:
NICU admissions and total number of days in NICU/baby | 2 months
number of patients hospitalized | at delivery
Total number of hospitalization days/ hospitalized participant | 2 months
Prevalence of gestational diabetes | up to delivery
Prevalence of preeclampsia | up to delivery
SNP | at delivery
  SNP analysis (genetic analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Eszter I Vanky, md phd, Study Director — Norwegian University of Science and Technology
Locations (13):
- Landspital University Hospital, Reykjavik, Iceland
- Norway (9):
  - Sykehuset Ålesund, Ålesund
  - Haukeland University Hospital, Bergen
  - Nordlandssykehuset HF, Bodø
  - Sykehuset Innlandet, Brumunddal
  - Vestre Viken Hospital Trust, Drammen
  - Vestre Viken Ringerike sykehus, Hønefoss
  - Sykehuset Telemark, Skien
  - St Olavs Hospital, Trondheim
  - Sentralsykehuset i Vestfold, Tønsberg
- Sweden (3):
  - Karolinska Universitetssjukhus, Stockholm
  - Norrlands universitetssjukhus, Umeå
  - Uppsala University Hospital, Uppsala

REFERENCES:
- [Result] Lovvik TS, Carlsen SM, Salvesen O, Steffensen B, Bixo M, Gomez-Real F, Lonnebotn M, Hestvold KV, Zabielska R, Hirschberg AL, Trouva A, Thorarinsdottir S, Hjelle S, Berg AH, Andrae F, Poromaa IS, Mohlin J, Underdal M, Vanky E. Use of metformin to treat pregnant women with polycystic ovary syndrome (PregMet2): a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2019 Apr;7(4):256-266. doi: 10.1016/S2213-8587(19)30002-6. Epub 2019 Feb 18. PMID 30792154
- [Derived] Ryssdal M, Skage JE, Jarmund AH, Hanem LGE, Lovvik TS, Giskeodegard GF, Iversen AC, Vanky E. Metformin Treatment in PCOS Pregnancies Reduces Maternal Infections and Increases the Risk of Allergies and Eczema in the Offspring: Post Hoc Analyses of Two Randomised Controlled Trials and One Follow-Up Study. BJOG. 2025 Nov;132(12):1823-1832. doi: 10.1111/1471-0528.18320. Epub 2025 Aug 11. PMID 40785326
- [Derived] Nordtvedt E, Kessler J, Ebbing C, Acharya G, Lovvik TS, Salvesen KA, Salvesen O, Vanky E, Kahrs BH. Placental and cerebral circulation in fetuses of mothers with polycystic ovary syndrome and the effect of Metformin exposure. BMC Pregnancy Childbirth. 2025 Jul 10;25(1):749. doi: 10.1186/s12884-025-07866-9. PMID 40640743
- [Derived] Husby AE, Simpson MR, Dalbye R, Larsen M, Vanky E, Lovvik TS. Childbirth experiences in women with polycystic ovary syndrome: A cohort study. Acta Obstet Gynecol Scand. 2024 Jun;103(6):1092-1100. doi: 10.1111/aogs.14800. Epub 2024 Feb 17. PMID 38366810
- [Derived] Stokkeland LMT, Giskeodegard GF, Ryssdal M, Jarmund AH, Steinkjer B, Madssen TS, Stafne SN, Stridsklev S, Lovvik TS, Iversen AC, Vanky E. Changes in Serum Cytokines Throughout Pregnancy in Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2022 Jan 1;107(1):39-52. doi: 10.1210/clinem/dgab684. PMID 34529073